CLINICAL TRIAL: NCT02219100
Title: Acceptability and Feasibility of a Demedicalized Medical Abortion Regimen in the Caucasus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1.2.3.1
Record Dates: First submitted 2014-07-29; First posted 2014-08-18 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Abortion, First Trimester
MeSH Terms: interventions — Mifepristone

ARMS (2):
- Home administration of mifepristone (Experimental): This arm consisted of women who chose home administration of 200 mg mifepristone.
  Interventions: Drug: Home administration of 200 mg mifepristone
- Clinic administration of mifepristone (No Intervention): This arm consisted of women who underwent clinic administration of 200 mg mifepristone.

INTERVENTIONS:
Drug: Home administration of 200 mg mifepristone — Home administration of 200 mg mifepristone
  Arms: Home administration of mifepristone

SUMMARY:
This study examined the acceptability and feasibility of using a simplified regimen of medical abortion in Armenia and Azerbaijan. It was hypothesized that home use of mifepristone and misoprostol, and buccal administration of misoprostol, would be both acceptable to women and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Good general health
* Living or working close to the study site
* Intrauterine pregnancy less than 64 days gestation
* Willing and able to sign consent forms
* Eligible for medical abortion according to the clinician's assessment
* Ready access to a telephone and emergency transportation
* Willing to provide an address and/or telephone number for purposes of follow-up
* Agree to comply with the study procedures and visit schedule

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
* IUD in place (IUD must be removed first)
* Chronic renal failure
* Concurrent long-term corticosteroid therapy
* History of allergy to mifepristone, misoprostol or other prostaglandin
* Hemorrhagic disorders or concurrent anticoagulant therapy
* Inherited porphyrias
* Other serious physical or mental health conditions

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 613 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Proportion of abortions that are complete without surgical intervention (unit: percent). | 15 days
  Percentage of women with complete abortion without the need of a surgical intervention.

SECONDARY OUTCOMES:
Proportion of women satisfied with procedure (unit: percent) and with side effects (unit: percent). | 15 days
  Woman's satisfaction with her medical abortion procedure and side effects experienced.

OTHER OUTCOMES:
Proportion of Women Who Select Home-use of Mifepristone | 1 week
Proportion of Women Who Select Home-use of Misoprostol | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Rena Bagirova, MD, Principal Investigator — Antenatal Clinic; Mehriban Huseynova, MD, Principal Investigator — Gynecology Department of the Central Regional Hospital; Aram Avalyan, MD, Principal Investigator — Vanadzor Hospital #1; Alla Minasyan, MD, Principal Investigator — Gyumri Maternity Hospital
Locations (5):
- Armenia (2):
  - Gyumri Maternity Hospital, Gyumri
  - Vanadzor Hospital #1, Vanadzor
- Azerbaijan (3):
  - Antenatal Clinic, Ganja
  - Family Planning Center, Ganja
  - Gynecology Department of the Central Regional Hospital, Zaqatala